CLINICAL TRIAL: NCT02392845
Title: A Pilot Dose Escalation Phase I Trial of a Densified Chemotherapy Association of Docetaxel and Epirubicin Driven by Mathematical Modeling in Metastatic Breast Cancer Patients: The MODEL1 Study
Brief Title: A Pilot Dose Escalation Trial of a Densified Chemotherapy Association of Docetaxel and Epirubicin Driven by Mathematical Modeling in Metastatic Breast Cancer Patients: The MODEL1 Study
Acronym: MODEL1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004.356
Record Dates: First submitted 2015-03-03; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Drug combination; Accelerated chemotherapy; Mathematical model; Hematotoxicity; Individualized dosage
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combination of Docetaxel (DTX) and Epirubicin (EPI) (Experimental)
  Interventions: Drug: Combination of Docetaxel (DTX) and Epirubicin (EPI)

INTERVENTIONS:
Drug: Combination of Docetaxel (DTX) and Epirubicin (EPI) — Six cycles of densified DTX+EPI chemotherapy (2 weeks per cycle) for each patient

SUMMARY:
To determine the maximum tolerated dose of a densified regimen of the association of docetaxel (DTX) and epirubicin (EPI), supported by the concomitant administration of hematopoietic growth factors in patients with metastatic breast cancer in first-line, optimizing in each patient the administration schedule using a formal procedure based on mathematical models in order to manage the severity of induced neutropenia.

The models used in this project allow:

* an optimal administration schedule of the planned total dose per cycle (number of infusions and calculating their rates and durations)
* an individualization of the administration schedule from the second cycle (based on observations from the first cycle), and
* an assessment of the risk of a dose-limiting toxicity event combining several severe non-hematological toxicities (conditioning the decision for dose escalation).

Using formal mathematical models the investigators expect controlling the hematological and non-hematological toxicities in order to realize the full series of six cycles of densified DTX+EPI chemotherapy (2 weeks per cycle) for each patient. For each patient, chemotherapy is considered feasible if it is possible, in the absence of tumor progression, to consider 6 cycles of treatment without observing any serious adverse events and without:

* patient death that may be related to the treatments;
* decision of the patient to interrupt treatment for physical or psychological tolerance reasons;
* decision of the investigator to discontinue treatment, in the absence of disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* ECOG performance status ≤ 2
* Diagnosed with metastatic HER2-negative hormone-resistant chemotherapy-naive breast cancers, previous adjuvant chemotherapy treatment are allowed.
* Histologically or cytologically proven breast cancer metastases or associated with CA 15-3 levels 50% above the normal value
* Hormone resistance defined by the presence of negative hormone receptors or disease progression within 6 months of the initiation of hormone therapy.
* Adequate renal and liver function (ASAT and ALAT < twice the upper limit normal value (ULN) if no liver metastases, or < 4×ULN if liver metastases; total bilirubin < 2×ULN),
* Adequate cardiac function (left ventricular ejection fraction (LVEF) > 50%),
* Neutrophils ≥ 1200/mm3
* Platelets ≥ 105/mm3

Exclusion Criteria:

* Cerebral metastases and meningeal involvement,
* Other malignant diseases,
* Significant comorbidities,
* Previous chemotherapy for metastatic disease, or previous chemotherapy with a total cumulative dose greater than 600 mg/m² for EPI or greater than 450 mg/m² for DTX

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Assessment of the risk of Dose-limiting Toxicities | 84 days (6 treatment cycles x 14 days)
  DLTs were defined as ≥ grade 3 vomiting, ≥ grade 3 mucositis,≥ grade 3 hand-foot syndrome (HFS), grade 2 vomiting plus grade 2 mucositis, or grade 2 vomiting plus grade 2 HFS

SECONDARY OUTCOMES:
Plasma concentration of Docetaxel and Epirubicin after administration | 84 days (6 treatment cycles x 14 days)
  Assessment of the pharmacokinetics of Docetaxel and Epirubicin
Tumor response for each patient with one or more measurable lesions | after 28 days (2 treatment cycles x 14 days) and 84 days (6 treatment cycles x 14 days)
  Measurement of tumor response by MRI for each patient with one or more measurable lesions, classified according to RECIST criteria
Progression-free survival | 115 days (study duration (6 treatment cycles x 14 days) + follow-up (31 days) when available)
Overall survival | 115 days (study duration (6 treatment cycles x 14 days) + follow-up (31 days) when available)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles FREYER, Professor, Principal Investigator — Hospices Civils de Lyon, Centre Hospitalier Lyon-Sud - Service d'oncologie médicale